CLINICAL TRIAL: NCT04822740
Title: Evaluation of the Use of a Continuous Glucose Monitoring System on Glycemic Equilibrium and Hypoglycemia in Diabetic Patients With Acute Coronary Syndrome Admitted in Intensive Care
Brief Title: Evaluation of Continuous Glucose Monitoring in Patients With ACS and Type 2 Diabetes in ICU
Acronym: EVASION
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: loss of equipment supplier
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP180484
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acute Coronary Syndrome; Type 2 Diabetes
Keywords: Acute coronary syndrome with ST-segment elevation; Acute coronary syndrome without ST-segment elevation; type 2 diabetes; Continuous glucose monitoring system (CGMS)
MeSH Terms: conditions — Acute Coronary Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel strategy (Experimental): Inserting the CGMS device with use of the results of the device in real time by the health care team
  * Insulin infusion according to the same local guidelines for insulin therapy in ACS
  * Transmission of real-time data to the nurse and use of the alarms of the device
  * Adaptation of insulin according to blood glucose measured by the CGMS device and according to the same protocol as the conventional arm
  * Glycemic range: maintain a blood glucose between 140 and 180 mg / dl
  Interventions: Device: Control Glucose Monitoring System
- Conventional strategy (Active Comparator): Inserting the CGMS device without the use of the results by the health care team: blinded CGMS (use of these results only at the end of the participation to analyze the main criterion)
  * Insulin infusion according to the same local guidelines for insulin therapy in ACS
  * Adaptation of insulin according to the capillary blood glucose levels performed every hourly if insulin dose change, every 2 hours if stable insulin dose according to local recommendations
  * Glycemic range: maintain a blood glucose between 140 and 180 mg / dl
  Interventions: Device: Control Glucose Monitoring System

INTERVENTIONS:
Device: Control Glucose Monitoring System — With a sensor, transmitter and display device (receiver and/or compatible smart device).
  The CGMS sends glucose readings to a compatible smart device every 5 minutes. In this study the CGMS for all patients with use of the results of the device in real time by the health care team for the Experimental arm and without the use of the results by the health care team for Active Comparator (Conventional strategy .

SUMMARY:
The investigators hypothesize that the use of a continuous glucose monitoring system (CGMS) can reduce glycemic variability assessed by coefficient of variation (CV) during the acute phase of acute coronary syndrome (ACS) in patients with diabetes treated by insulin infusion.

The purpose of this project is to assess the impact of the use of CGMS on glycemic variability in diabetic patients with ACS .

This is a randomized, multicenter (2 centers), open study. The patients included, as soon as possible, after admission will be randomized before the beginning of insulin therapy with intravenous insulin .

DETAILED DESCRIPTION:
The aim of this study is to assess the impact of the use of a continuous glucose monitoring system (CGMS) on glycemic variability in diabetic patients admitted in Intensive care unit (ICU) for an acute coronary syndrome ( ST Segment Elevation Myocardial Infarction (STEMI) or Non-ST segment elevation myocardial infarction (NSTEMI)) and treated with insulin infusion with a standardized protocol.

60 patients in 2 centers will be included, and all patient will have the CGMS.

Randomization will be done in the 12 hours after admission. Participants will be randomized in two groups :

* Conventional strategy: management of hyperglycemia with standard of care, glycemia monitoring with capillary blood glucose measurement. The goal is to maintain glycemia between 140-180mg/dL. CGMS will be blinded in this group.
* Novel strategy: management of hyperglycemia using CGMS. Measurements of CGMS will be transmitted in real time to medical staff and use to maintain glycemia between 140-180mg/dL. Alarms will be set to warn medical staff in case of glycemia outside the range.

The duration of follow-up for each patient will be 72 hours or until discharge from Intensive care unit (if <72 hours)

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years old admitted to Cardiac Intensive Care Unit (CICU for acute coronary syndrome (ACS):

   * ACS with STsegment elevation (STEMI), defined by thoracic pain of more than 30 minutes and sus-offset persist of the ST segment at ECG in two contiguous derivations.
   * ACS without ST segment elevation (NSTEMI), defined by a significant elevation of the troponin (> 99th percentile) with one of the following signs:

     * Symptoms of ischemia
     * Recent modification of the ST or wave segment T to ECG
     * Appearance of a wave q at ECG
     * Loss of segmental viability of myocardial imaging
     * intracoronal thrombus in angiography
2. patient with type 2 diabetes (defined according to the American Diabetes Association (ADA) recommendations) known with:

   * be a hyperglycemia> 180 mg / dl to admission that requires intravenous insulin therapy
   * Either chronic insulin treatment before admission
3. Patient who has not yet received insulin therapy with intravenous insulin since admission
4. Signed informed consent
5. oral and written comprehension of the French language

Exclusion Criteria:

1. Patient with hemodynamic instability (shock, catecholamine use, mechanical ventilation, circulatory assistance ...)
2. Patient admitted to the CICU since more than 24 hours
3. Patient requiring Corticotherapy
4. patient with type 1 diabetes (defined according to the ADA recommendations)
5. Needs to perform MRI during CICU stay
6. Pregnancy or breastfeeding
7. patient under legal protection
8. Patient with no social security
9. Patient participating in another interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Glycemic variability by the coefficient of variation of blood glucose in percent | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Glycemic variability assessed by the coefficient of variation of blood glucose in percent ((standard deviation / medium blood glucose) x 100)

SECONDARY OUTCOMES:
Glycemic variability measured by MAGE index | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Glycemic variability measured by MAGE index (Mean Amplitude of Glycemic Excursions Index)
Glycemic variability measured by LBGI | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Glycemic variability measured by LBGI ( (Low Blood Glucose Index)
Glycemic variability measured by standard deviation | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Glycemic variability measured by standard deviation of blood glucose
Number of symptomatic hypoglycemia | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Number of symptomatic hypoglycemia in both groups.
Number of hypoglycemia during ICU stay | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Number of hypoglycemia (<54, <70 and < 90 mg/dl) during ICU stay in both groups.
Time spent in glycemic target, in hypoglycemia, and in hyperglycemia | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Time spent in glycemic target (140-180 mg/dl), in hypoglycemia <50 and < 90 mg/dl), and in hyperglycemia (>180/250 mg/dl)
Mean insulin perfusion rate | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Mean insulin perfusion rate (Total insulin dose per total time)
Failure of CGMS failure | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Failure of CGMS failure (no or incomplete glucose data)
Local complications of GGMS | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Local complications of GGMS: bleeding with CGM withdrawn, cutaneous intolerance, CGM withdrawn
Usefulness for nurse | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Usefulness for nurse (survey)
Patient satisfaction | From enrollment to the first 72 hours of hospitalization or until discharge of ICU (if <72 hours).
  Patient satisfaction (satisfaction questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre RIVELINE, pr, Study Director — APHP
Locations (1):
- Lariboisière Hospital, Paris, Île-de-France Region, France